CLINICAL TRIAL: NCT02945618
Title: Neurocryostimulation for the Treatment of Acute Lateral Ankle Sprain : a Single Blind Randomized Controlled Trial
Brief Title: Neurocryostimulation for Acute Lateral Ankle Sprain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean-Sébastien Roy, Associate Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cryofos
Record Dates: First submitted 2016-10-23; First posted 2016-10-26 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Ankle Sprain
Keywords: cryotherapy; physical therapy
MeSH Terms: conditions — Ankle Injuries | interventions — Ice

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neurocryostimulation (Experimental): CRYOFOS will be applied on the ankle at the end of each of the 8 sessions (in accordance to the protocol established). The treatment time with the CRYOFOS will take between 1 and 2 minutes, and will be pain-free.
  Both groups will also receive the same conventional program consisting of: compression, bracing, early mobilization (including manual therapy), strengthening (isometric and isotonic using elastic bands) and proprioception (using proprioception boards) exercises, according to the grade of the sprain and the stage of biological ligament healing.
  Interventions: Device: Neurocryostimulation
- Conventional program with ice (Active Comparator): The control group will receive the same conventional program (as the experimental group) consisting of: compression, bracing, early mobilization (including manual therapy), strengthening (isometric and isotonic using elastic bands) and proprioception (using proprioception boards) exercises, according to the grade of the sprain and the stage of biological ligament healing. Ice will be applied to the ankle for 15 minutes at the end of each of the 8 sessions.
  Interventions: Other: Ice

INTERVENTIONS:
Device: Neurocryostimulation — CRYOFOS will be applied on the ankle at the end of each of the 8 sessions (in accordance to the protocol established). The treatment time with the CRYOFOS will take between 1 and 2 minutes, and will be pain-free.
  Both groups will also receive the same conventional program consisting of: compression, bracing, early mobilization (including manual therapy), strengthening (isometric and isotonic using elastic bands) and proprioception (using proprioception boards) exercises, according to the grade of the sprain and the stage of biological ligament healing.
  Other Names: Hyperbaric gazeous cryotherapy; Cryostimulation
  Arms: Neurocryostimulation
Other: Ice — The control group will receive the same conventional program (as the experimental group) consisting of: compression, bracing, early mobilization (including manual therapy), strengthening (isometric and isotonic using elastic bands) and proprioception (using proprioception boards) exercises, according to the grade of the sprain and the stage of biological ligament healing. Ice will be applied to the ankle for 15 minutes at the end of each of the 8 sessions.
  Other Names: Conventional program with ice
  Arms: Conventional program with ice

SUMMARY:
The objective of this exploratory randomized control trial is to compare, in participants with acute lateral ankle sprain (LAS) , the reduction of symptoms and functional limitations between two groups of subjects who undergo a conventional rehabilitation program with (experimental group) or without CRYOFOS (comparison group). The hypothesis is that CRYOFOS will lead to a faster reduction of symptoms and functional limitations, and a faster return to daily living activities.Thirty-six participants of 18 years of age and older with acute LAS (sustained a LAS three days or less before the first evaluation session) will be recruited and randomly assigned to either a group receiving conventional rehabilitation program with the addition of CRYOFOS (experimental group; n=18), or to a group only receiving the conventional rehabilitation program (comparison group; n=18). This single-blind (evaluator), parallel-group RCT will include five evaluation sessions over 6 weeks (baseline, day 7, week 2, week 4 and week 6) and 8 treatment sessions (1st and 2nd weeks: 3 sessions/week; 3rd and 4th weeks: 1 session/week) during a 4-week period. The primary outcome will be the functional limitations, evaluated using the Lower Extremity Functional Scale (LEFS).

DETAILED DESCRIPTION:
Lateral ankle sprain (LAS) is one of the most common reasons for primary care office and emergency department visits, with an overall incidence of 2.15 per 1,000 person-years in the United States.In its acute phase, LAS is associated with swelling, haematoma and pain over the anterior talofibular and calcaneofibular ligaments, as well as ligamentous laxity of these ligaments. Interventions following acute LAS are based upon the three stages of biological ligament healing: inflammatory phase, proliferation phase (6 weeks to 3 months after trauma) and remodelling or maturation phase (until 1 year after trauma). The initial treatment during inflammatory phase is directed towards avoiding or diminishing excess swelling and ongoing injury, thus optimizing the healing process. Therefore, RICE (Rest, Ice [cryotherapy], Compression, Elevation) is the treatment of choice for the first 7 to 10 days to reduce pain and swelling. Cryotherapy has been used for a long time in rehabilitation; mainly using ice, cool packs or cold water. Lately, a new device, the CRYOFOS, has been developed to provide more performing ways to use cryotherapy. CRYOFOS uses a fluid (hyperbaric CO²) that is sprayed in the form of dry ice on the body region to be treated. It leads to a so-called thermal shock, which sees the skin temperature cooled from 32 ˚C to 2-4 ˚C in 30 sec.While CRYOFOS seems, theoretically, better than other cooling procedures, its superiority has never been determined following acute injuries such as LAS. Considering the extensive use of cold in the management of acute LAS, it would be even more relevant to examine the impact of cryotherapy on both the reduction of symptoms and the functional limitations of subjects who sustained a LAS.

The objective of this exploratory randomized control trial is to compare, in participants with acute lateral ankle sprain (LAS) , the reduction of symptoms and functional limitations between two groups of subjects who undergo a conventional rehabilitation program with (experimental group) or without CRYOFOS (comparison group). The hypothesis is that CRYOFOS will lead to a faster reduction of symptoms and functional limitations, and a faster return to daily living activities.Thirty-six participants of 18 years of age and older with acute LAS (sustained a LAS three days or less before the first evaluation session) will be recruited and randomly assigned to either a group receiving conventional rehabilitation program with the addition of CRYOFOS (experimental group; n=18), or to a group only receiving the conventional rehabilitation program (comparison group; n=18). This single-blind (evaluator), parallel-group RCT will include five evaluation sessions over 6 weeks (baseline, day 7, week 2, week 4 and week 6) and 8 treatment sessions (1st and 2nd weeks: 3 sessions/week; 3rd and 4th weeks: 1 session/week) during a 4-week period. The primary outcome will be the functional limitations, evaluated using the Lower Extremity Functional Scale (LEFS). Secondary outcomes will include the level of ankle pain, evaluated using Numeric Pain Rating Scales (NPRS), weight-bearing ankle dorsiflexion range of motion (also called Bent Knee DorsiFlexion test), assessed with the maximal advancement of the tibia over the talus in a weight-bearing position, and joint swelling, using the Figure-of-Eight method.

Both groups will receive the same conventional program consisting of: compression, bracing, early mobilization (including manual therapy), strengthening (isometric and isotonic using elastic bands) and proprioception (using proprioception boards) exercises, according to the grade of the sprain and the stage of biological ligament healing. However, for the experimental group, CRYOFOS will be applied on the ankle at the end of each of the 8 sessions (in accordance to the protocol established).

Descriptive statistics will be used for all outcome measures at each measurement time to summarise results. Baseline demographic data will be compared (independent t-test and Chi-squared tests) to establish the comparability of groups. All data will be tested to check the distributional assumptions for the inferential statistical analyses. An intention-to-treat analysis will be used in which all participants will be analysed in the group to which they were originally assigned. All dropouts and the reason for dropping out of the study will be reported. Any harm or unintended effects during the programs will be recorded. A 2-way ANOVA (2 cryotherapy [CRYOFOS or Ice] x 5 Time [baseline, day 7, week 2, week 4, week 6]) will be used to analyse the effects of CRYOFOS on primary outcome (LEFS) and secondary outcomes (SPSS 22, proc GENLIN [Generalized Estimating Equations for repeated measures]).

ELIGIBILITY:
Inclusion Criteria:

* LAS three days or less before the first evaluation session
* presence of a lateral hematoma and swelling
* tenderness at the anterior lateral ligament without or with anterior drawer instability

Exclusion Criteria:

* present a bony ankle injury (indicated by Ottawa ankle rules)
* had sustained a similar injury of the same joint within the last 6 months
* require bed rest, hospitalisation, casting or surgery
* had a previous fracture of the same ankle
* signs or symptoms of a previous injury at any of the other joints of the lower limbs or trunk
* contraindication to cryotherapy including cryoglobulinemia, peripheral vascular disease or Raynaud's syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in lower limb functional level at 6 weeks | Baseline-6 weeks
  Lower Extremity Functional Scale (LEFS), an auto-administered questionnaire of functional capacity

SECONDARY OUTCOMES:
Change from Baseline in pain level at 6 weeks | Baseline-6 weeks
  Visual analog scale for pain
Change from Baseline in pain level at 1 week | Baseline-1 week
  Visual analog scale for pain
Change from Baseline in pain level at 2 weeks | Baseline-2 weeks
  Visual analog scale for pain
Change from Baseline in pain level at 4 weeks | Baseline-4 weeks
  Visual analog scale for pain
Change from Baseline in ankle oedema at 6 weeks | Baseline-6 weeks
  Figure-of-eight for ankle oedema
Change from Baseline in ankle oedema at 4 weeks | Baseline-4 weeks
  Figure-of-eight for ankle oedema
Change from Baseline in ankle oedema at 2 weeks | Baseline-2 weeks
  Figure-of-eight for ankle oedema
Change from Baseline in ankle oedema at 1 week | Baseline-1 week
  Figure-of-eight for ankle oedema
Change from Baseline in dorsiflexion range of motion at 6 weeks | Baseline-6 weeks
  Hallux-to-wall distance for dorsiflexion range of motion
Change from Baseline in dorsiflexion range of motion at 1 week | Baseline-1 week
  Hallux-to-wall distance for dorsiflexion range of motion
Change from Baseline in dorsiflexion range of motion at 2 weeks | Baseline-2 weeks
  Hallux-to-wall distance for dorsiflexion range of motion
Change from Baseline in dorsiflexion range of motion at 4 weeks | Baseline-4 weeks
  Hallux-to-wall distance for dorsiflexion range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sebastien Roy, PhD, Principal Investigator — Universite Laval
Locations (1):
- Laval University, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tittley J, Hebert LJ, Roy JS. Should ice application be replaced with neurocryostimulation for the treatment of acute lateral ankle sprains? A randomized clinical trial. J Foot Ankle Res. 2020 Dec 1;13(1):69. doi: 10.1186/s13047-020-00436-6. PMID 33261633